CLINICAL TRIAL: NCT05213247
Title: A Short-Term Follow-Up Study on the Effect of Khat Chewing on Blood Pressure and Heart Rate Among Healthy Adults in Taiz, Yemen: Its Associated Factors and SDS-Khat
Brief Title: Effect of Khat Chewing on Blood Pressure and Heart Rate Among Healthy Adults
Status: Completed | Type: Observational
Sponsor: Aljanad University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mujeeb Abdullah Saeed Sultan, Head of Pharmacy Department, Aljanad University for Science and Technology
Other Study IDs: JustMed01/2021
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Blood Pressure; Heart Rate
Keywords: Khat-SDS; Blood Pressure; Heart Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: electronic apparatus (visocor OM50). — Measurement of blood pressure and heart rate

SUMMARY:
This study is a cross sectional study

DETAILED DESCRIPTION:
Objective: This study aims to investigate .ht short-term effect of khat on the diastolic and systolic blood pressure (DBP, SBP) and heart rate (HR) of yemeni adults. Factors associated with Khat chewing and Khat-dependence were also investigated. That the khat chewing is a growing public habit among yemeni people.

ELIGIBILITY:
The participant should be free of any disease and should avoid eating or drinking anything that could affect on BP and HR within two khat before hours chewing (zero time)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a cross-sectional study conducted from April to September 2021 in Taiz, Yemen. 100 healthy adults were selected using a random sampling method.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | April- December 2021
  Elevation of blood pressure due to khat Chewing

CONTACTS AND LOCATIONS:
Overall Officials: Mujeeb Sultan, Principal Investigator — Aljanad University for Science and Technology
Locations (1):
- Mujeeb Sultan, Ta‘izz, Yemen

IPD SHARING:
Plan to Share IPD: No